CLINICAL TRIAL: NCT02028624
Title: Lifestyle Interventions Based on the Mediterranean Diet for Patients With Rheumatoid Arthritis: a Randomized Controlled Trial
Brief Title: Lifestyle Interventions Based on the Mediterranean Diet for Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: State Scholarships Foundation, Athens, Greece (Unknown)
Responsible Party: Principal Investigator, M. Yannakoulia, Dr Mary Yannakoulia, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RASt
Record Dates: First submitted 2014-01-01; First posted 2014-01-07 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Mediterranean diet; Lifestyle intervention; Adiponectin; Telephone counseling
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Face-to-face (Experimental): Patients received face-to-face nutrition counseling.
  Interventions: Behavioral: Nutrition counseling
- Telephone (Experimental): Patients received telephone nutrition counseling.
  Interventions: Behavioral: Nutrition counseling
- Minimum Intervention (No Intervention): Patients in this group received no further lifestyle-related counseling and contact until the 6-month evaluation.

INTERVENTIONS:
Behavioral: Nutrition counseling — Patients received nutrition counseling, through one-to-one sessions conducted once a month, until the 6-month evaluation. Nutrition counseling was based on goal-setting and aimed at increasing adherence to Mediterannean diet.
  Arms: Face-to-face; Telephone

SUMMARY:
Aim of the present study was to evaluate the effect of different lifestyle intervention administrations, in increasing adherence to the Mediterranean diet in a group of patients with RA living in the Mediterranean basin, and, thus, in improving parameters related to subjective and objective disease markers, including plasma adiponectin concentrations.

DETAILED DESCRIPTION:
The effect of various dietary regimens and nutrient supplementation on rheumatoid arthritis (RA) has been previously explored, with the majority of the evidence supporting the beneficial effect of n-3 polyunsaturated fatty acids (PUFAs), consumed mainly as fish oil supplements. However, many capsules should be taken on a daily basis (10 - 15) in order to improve health status, increasing, thus, the high drug burden these patients may encounter; inability to comply with supplementation, as depicted in drop-out rates and adverse reactions, is also of concern. On the other hand, the so far investigation of specific dietary patterns, namely elemental or vegetarian diets, revealed similar limitations regarding inability to comply, without producing clear benefit.

The last decade, a traditional dietary pattern, the Mediterranean diet, has also been investigated in patients with RA. This pattern is characterized by abundance of plant foods (fruits, mainly as typical daily desserts, vegetables, bread, other forms of cereals, beans, nuts, and seeds), olive oil as the principal source of fat, moderate amounts of dairy products (mainly cheese and yogurt), low to moderate amounts of fish and poultry, red meat in low amounts and wine consumed in moderation, normally with meals. Adherence to the Mediterranean diet has been associated with a significant reduction in total mortality and improvement in longevity, as well as with lower incidence of atherosclerosis, coronary heart disease, metabolic syndrome and biochemical markers related to insulin resistance and inflammation. In RA, in specific, it has been shown to improve objective and subjective measures. It is also worth mentioning that this type of intervention produced negligible or no adverse effects or drop-out in RA patients. However, it has been implemented in North-European populations with a background diet far away from the Mediterranean dietary habits. It would be interesting to study the effect of a Mediterranean diet-based intervention in a Mediterranean population of RA patients, evaluate their adherence and changes in subjective disease measures as well as in biochemical markers. One of the markers of interest is adiponectin, a large 30-kDa protein produced mainly by adipocytes, sharing strong homologies with TNF and the complement factor C1q. Plasma levels of adiponectin have been negatively associated with indices of obesity, insulin resistance and cardiovascular disease. However, its role in RA is still controversial with some evidence indicating a proinflammatory effect and some other suggesting antiinflammatory properties of this adipocytokine.

Aim of the present study was to evaluate the effect of different lifestyle intervention administrations, in increasing adherence to the Mediterranean diet in a group of patients with RA living in the Mediterranean basin, and, thus, in improving parameters related to subjective and objective disease markers, including plasma adiponectin concentrations.

ELIGIBILITY:
Inclusion Criteria:

* adults
* rheumatoid arthritis diagnosis according to the 1987 criteria of the American College of Rheumatology
* clinically non active disease, as assessed and documented by the patient's own rheumatology specialist

Exclusion Criteria:

* being on a slimming or any other special diet during the previous year, or being diagnosed with other serious medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline Mediterranean Diet Score at 6 months | 6 months
Change from baseline Disease Activity Score (DAS28) at 6 months | 6 months
Change from baseline Health Assessment Questionnaire (HAQ) Score at 6 months | 6 months
Change from baseline Short Form-36 Health Survey (SF-36) score at 6 months | 6 months
Change from baseline energy intake at 6 months | 6 months
Change from baseline in macronutrients intake at 6 months | 6 months
Age | baseline
Height | baseline
Change from baseline body weight at 6 months | 6 months
Change from baseline systolic blood pressure at 6 months | 6 months
Change from baseline plasma adiponectin concentrations at 6 months | 6 months
Change from baseline plasma glucose levels at 6 months | 6 months
Change from baseline serum triglycerides levels at 6 months | 6 months
Change from baseline plasma HDL-cholesterol levels at 6 months | 6 months
Years of education | baseline
Change from baseline diastolic blood pressure at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Yannakoulia, PhD, Study Director — Harokopio University
Locations (2):
- Greece (2):
  - Euroclinic Private Hopsital, Athens
  - Laiko General Hospital, Athens